CLINICAL TRIAL: NCT03940391
Title: Effect of an Adjunctive Sedative for the Patients With Histories of Paradoxical Reaction to Midazolam During Sedative Endoscopy
Brief Title: Effect of the Antihistamine Injection to Prevent Paradoxical Reaction During Sedative Endoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Su Jin Chung, Professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H-1093-054-1017
Record Dates: First submitted 2019-04-24; First posted 2019-05-07 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Endoscopy
Keywords: paradoxical reaction; midazolam
MeSH Terms: interventions — Chlorpheniramine; Midazolam

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- antihistamine combination (Experimental): Participants in this group will get combination chlorpheniramine and midazolam injection for sedative endoscopy.
  Interventions: Drug: Chlorpheniramine and midazolam
- midazolam (Placebo Comparator): Participants in this group will get only midazolam injection for sedative endoscopy
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Chlorpheniramine and midazolam — Administration of chlorpheniramine injection as an adjunctive sedative during sedative endoscopy.
  Arms: antihistamine combination
Drug: Midazolam — Administration of midazolam as a sedative during sedative endoscopy as routine clinical practice.
  Arms: midazolam

SUMMARY:
This single-blind prospective study is aimed to investigate the effect of antihistamine as an adjunctive sedative for the patients with histories of severe paradoxical reaction to midazolam during sedative endoscopy. Participating patients are to receive antihistamine intravenously in addition to midazolam. The primary outcome is the reduction of paradoxical reaction in the antihistamine combination group. The secondary outcome is to compare sedation quality, performance quality, reduction of total midazolam dose will be analyzed between antihistamine combination and midazolam only group.

DETAILED DESCRIPTION:
The present study will be conducted at Seoul National University Hospital Gangnam center between May 2019 and April 2020. Participants who have histories of paradoxical reaction to sedative endoscopy in medical record gave consent on the day of the endoscopy and were assigned to receive the combination of chlorpheniramine (4-6mg) with midazolam(1-10mg) Meanwhile, the patients do not want the use of chlorpheniramine and were assigned to midazolam alone as routine clinical practice. Research medication (chlorpheniramine) was administered 2 to 3 minutes before the administration of midazolam outside of endoscopy room. The blinded endoscopist and assistant nurse are going to perform induction for moderate sedation using incremental doses of the intravenous midazolam (1-2 mg) given every 2 minutes. The endoscopists and assistant nurses will assess the occurrence of severe paradoxical reaction (Grade 3) and other major quality outcomes (procedure/intubation time, sedation quality, completeness of procedure [10 Key image documentation], the satisfaction of procedure, side effects). The endoscopists and nurses will individually rate outcome measure using a 5-point Likert scale.

ELIGIBILITY:
Inclusion Criteria:

* Previous histories of the paradoxical reaction during a sedative endoscopic examination

Exclusion Criteria:

* inability to execute informed consent
* allergic to antihistamine agent
* pregnancy
* severe cardiopulmonary disease
* prior administration of antihistamine on the same day

Ages: 19 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-04-14 (Estimated); Study Completion 2020-04-14 (Estimated)

PRIMARY OUTCOMES:
Occurrence of severe paradoxical reaction (>= level 3) | 1 day
  (1) irrational talking or increased talkativeness such as mumbling to himself/herself; (2) restlessness or loss of cooperation such as resisting the insertion of endoscope or trying to bite the scope; (3) excessive movement requiring repositioning such as jerking or swinging movements of the arms and legs or trying to draw out the scope or mouthpiece; and (4) hostile action such as trying to strike the endoscopists or attending nurses.

SECONDARY OUTCOMES:
procedure/intubation time | 1 day
  procedural time (time from scope insertion to scope out) Intubation time (time from scope insertion to upper esophagus)
Dose of midazolam | 1 day
  total amount of benzodiazepine
completeness of procedure | 1 day
  photo documentation of key anatomical area
Satisfaction for Quality of sedation | 1 day
  5-point Likert scale : endoscopists and assistant nurses
  1. Strongly unsatisfied
  2. Unsatisfied
  3. Neither satisfied nor unsatisfied
  4. Satisfied
  5. Strongly satisfied
Satisfaction for the procedure | 1 day
  5-point Likert scale for pain and sedation: patients
  1. Strongly unsatisfied
  2. Unsatisfied
  3. Neither satisfied nor unsatisfied
  4. Satisfied
  5. Strongly satisfied
adverse events | 1 day
  hypoxia, arrythmia, low blood pressure and administration of antidote

CONTACTS AND LOCATIONS:
Locations (1):
- Healthcare System Gangnam Center, Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sachar H, Pichetshote N, Nandigam K, Vaidya K, Laine L. Continued midazolam versus diphenhydramine in difficult-to-sedate patients: a randomized double-blind trial. Gastrointest Endosc. 2018 May;87(5):1297-1303. doi: 10.1016/j.gie.2017.01.028. Epub 2017 Jan 31. PMID 28159539
- [Result] Nusrat S, Madhoun MF, Tierney WM. Use of diphenhydramine as an adjunctive sedative for colonoscopy in patients on chronic opioid therapy: a randomized controlled trial. Gastrointest Endosc. 2018 Oct;88(4):695-702. doi: 10.1016/j.gie.2018.04.2342. Epub 2018 Apr 22. PMID 29689257
- [Result] Tae CH, Kang KJ, Min BH, Ahn JH, Kim S, Lee JH, Rhee PL, Kim JJ. Paradoxical reaction to midazolam in patients undergoing endoscopy under sedation: Incidence, risk factors and the effect of flumazenil. Dig Liver Dis. 2014 Aug;46(8):710-5. doi: 10.1016/j.dld.2014.04.007. Epub 2014 Jun 2. PMID 24893689
- [Result] Tu RH, Grewall P, Leung JW, Suryaprasad AG, Sheykhzadeh PI, Doan C, Garcia JC, Zhang N, Prindiville T, Mann S, Trudeau W. Diphenhydramine as an adjunct to sedation for colonoscopy: a double-blind randomized, placebo-controlled study. Gastrointest Endosc. 2006 Jan;63(1):87-94. doi: 10.1016/j.gie.2005.08.015. PMID 16377322